CLINICAL TRIAL: NCT00963924
Title: A Placebo-controlled Trial of D-cycloserine Augmentation of Cognitive Remediation in Schizophrenia
Brief Title: D-cycloserine Augmentation of Cognitive Remediation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Donald C. Goff, MD, Director of the Schizophrenia Clinical and Research Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008P002237; 5P50MH060450 (NIH); DATR A3-NSC
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Schizophrenia
Keywords: Cognitive Impairment; Neuroplasticity; D-cycloserine; NMDA; Anti-Bacterial Agents; Mental Disorders; Psychotic Disorders; Antitubercular Agents; Schizophrenia and Disorders with Psychotic Features; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Cognitive Dysfunction; Mental Disorders; Psychotic Disorders; Schizophrenia Spectrum and Other Psychotic Disorders | interventions — Cycloserine; Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- D-cycloserine (Experimental): Participants will receive D-cycloserine weekly, one hour before the first cognitive remediation session of the week, for eight weeks.
  Interventions: Drug: D-cycloserine; Behavioral: Cognitive Remediation
- Placebo (Placebo Comparator): Participants will receive placebo weekly, one hour before the first cognitive remediation session of the week, for eight weeks.
  Interventions: Drug: Placebo; Behavioral: Cognitive Remediation

INTERVENTIONS:
Drug: D-cycloserine — 50 mg by mouth one hour before first cognitive remediation session each week for eight weeks.
  Other Names: Cycloserine
  Arms: D-cycloserine
Drug: Placebo — Placebo by mouth one hour before first cognitive remediation session each week for eight weeks.
  Arms: Placebo
Behavioral: Cognitive Remediation — 40 one-hour daily sessions of cognitive remediation (Brain Fitness Program) over eight weeks.
  Other Names: Brain Fitness Program

SUMMARY:
This study seeks to examine the effects of D-cycloserine augmentation on cognitive remediation for patients diagnosed with schizophrenia. We will test the hypotheses that D-cycloserine will significantly improve cognitive performance, negative symptoms, and measures of functioning compared to placebo when combined with eight weeks of cognitive remediation. We expect that these effects will persist when assessed at six-month follow up.

DETAILED DESCRIPTION:
D-cycloserine has been shown to enhance learning in animal models and, in a previous trial, once-weekly D-cycloserine improved negative symptoms in schizophrenia subjects. We set out to test whether DCS combined with cognitive remediation would improve learning of a practiced auditory discrimination task and whether gains would generalize to unpracticed cognitive tasks.

The proposed study consists of an 8-week, placebo-controlled, double-blind, parallel-group trial of D-cycloserine augmentation of cognitive remediation in schizophrenia outpatients. The primary outcome measure is change in performance on the MATRICS cognitive battery composite score after 8 weeks. Secondary outcome measures include a measure of processing speed assessed after weeks 1, 2, 4 & 8, and changes in negative symptoms and measures of functioning after 4 and 8 weeks. In addition, all outcome measures will be repeated at 6 months to assess persistence of benefit.

Hypotheses:

1. D-cycloserine will significantly improve cognitive performance as measured by the composite score on the MATRICS battery compared to placebo after 8 weeks of cognitive remediation.
2. D-cycloserine will significantly improve negative symptoms as measured by the SANS compared to placebo after 8 weeks when combined with cognitive remediation.
3. D-cycloserine will significantly improve measures of functioning (GAS, QoL and CGI) at 8 weeks compared to placebo when combined with cognitive remediation.
4. D-cycloserine effects on cognition, negative symptoms and functioning will persist compared to placebo when assessed at 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-65 years
* Diagnosis of schizophrenia or schizoaffective disorder, depressed type
* Stable dose of antipsychotic for at least 4 weeks
* Able to provide informed consent
* Able to complete a cognitive battery
* Able to perform the cognitive remediation exercises

Exclusion Criteria:

* Current treatment with clozapine
* Dementia
* Seizure disorder
* Unstable medical illness
* Renal insufficiency measured as eGFR >60mg/dL/min
* Active substance abuse: positive urine toxic screen
* Pregnancy, nursing, or unwilling to use appropriate birth control measures during participation if female and fertile.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald C. Goff, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Cain CK, McCue M, Bello I, Creedon T, Tang DI, Laska E, Goff DC. d-Cycloserine augmentation of cognitive remediation in schizophrenia. Schizophr Res. 2014 Mar;153(1-3):177-83. doi: 10.1016/j.schres.2014.01.016. Epub 2014 Jan 30. PMID 24485587

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 54 patients were assessed for eligibility; however, 14 were excluded (11 were ineligible, and 3 withdrew consent). 40 participants were randomized, however 4 were excluded (1 serious adverse event, 2 withdrew consent, and 1 was lost to follow up), therefore 36 entered the treatment phase.
Period: Overall Study
Arm/Group | D-cycloserine | Placebo
Started | 18 | 18
Completed | 17 | 15
Not Completed | 1 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Changed antipsychotic | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-cycloserine | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 18 | 36
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.5) | 46.2 (13.3) | 47.5 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 16 | 15 | 31
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS)
Description: Change of a composite score from baseline to week 8 on the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS). The MATRICS consists of 10 cognitive tasks that are used to calculate scores in 7 cognitive domains: speed of processing, attention/vigilance, working memory, verbal learning, visual learning, reasoning and problem solving, and social cognition. The raw scores on each cognitive task are transformed on a normative scale into t-scores, and then these scores are combined to calculate the domain scores. The composite score is calculated by averaging all domain t-scores to come up with one overall cognitive composite t-score. For all scores on the assessment, the higher the score the better the performance on the task.
Time Frame: Baseline vs. Week 8
Population: 18 participants in each arm had baseline values available for analysis. 17 in the D-cycloserine arm and 15 in the placebo arm had week 8 values available for analysis.
Measure: Mean (Standard Deviation); unit: t-scores
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
t-scores
  Baseline | 32.1 (13.4) | 33.0 (13.8)
  Week 8: number analyzed (Participants) | 17 | 15
  Week 8 | 32.24 (13.53) | 33.8 (14.50)

2. Primary Outcome: Scale for Assessment of Negative Symptoms (SANS)
Description: The total scores from baseline and week 8 on the scale for the assessment of negative symptoms (SANS) total score. Total SANS scores range from 0-100. The SANS is comprised of 5 subscores: Affective Flattening or Blunting (score range 0-35), Alogia (score range 0-20), Avolition-Apathy (score range 0-15), Anhedonia-Asociality (score range 0-20), and Attention (0-10). For each scale, the higher the score the more prominent the negative symptoms were. The total score was computed by adding all the sub-scale total scores. Scores are reported for baseline and week 8.
Time Frame: Baseline vs. Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 24.6 (13.5) | 25.8 (10.7)
  Week 8: number analyzed (Participants) | 17 | 15
  Week 8 | 22.41 (10.28) | 24.67 (10.42)

3. Primary Outcome: Auditory Discrimination Task: Interstimulus Interval (ISI)
Description: The auditory discrimination task involved trials in which the subject differentiated between rapidly-presented frequency-modulated sweeps separated by a short interstimulus interval (ISI). In this task, sustained successful performance is more difficult with shorter stimulus presentations and ISIs (which were equal within a trial). Thus, our dependent measure was the shortest stimulus duration/ISI, in ms, for trials in which subjects were able to perform the task at 85% accuracy, referred to as ISI for simplicity. The shorter the score the better the performance on the task. Scores are reported for baseline and week 8.
Time Frame: Baseline vs. Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
milliseconds
  Baseline | 163.5 (86.5) | 124.8 (93.0)
  Week 8: number analyzed (Participants) | 17 | 15
  Week 8 | 91.7 (65.4) | 127.9 (115.6)

4. Secondary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The baseline score on the positive symptom sub-scale of the Positive and Negative Syndrome Scale (PANSS). Total PANSS positive symptom sub-scale scores range from 7-49. The PANSS positive symptom sub-scale is comprised of 7 items rated on a scale of 1-7: delusions, conceptual disorganization, hallucinatory behavior, excitement, grandiosity, suspiciousness/persecution, and hostility. A score of one on each item 1 absent, 2 is minimal, 3 is mild, 4 is moderate, 5 is moderately severe, 6 is severe, and 7 is extreme. The total score was computed by adding all the items on the sub-scale together. The higher a score the more prominent a positive symptom is.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale | 61.8 (11.4) | 64.1 (15.5)

5. Secondary Outcome: Global Assessment of Functioning Scale (GAS)
Description: The Global Assessment of Functioning Scale (GAS) measured at baseline. This scale measures social, occupational, and psychological functioning, on a scale of 0-100. The higher the score, the greater a participant's functioning level.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale | 53.7 (6.5) | 50.8 (11.2)

6. Secondary Outcome: Heinrich Quality of Life Scale (QoL)
Description: Baseline scores of the Heinrich Quality of Life Scale, a 21 item scale designed and validated to measure intrapsychic foundations, interpersonal relations, instrumental role, and common objects and activities in patients diagnosed with Schizophrenia. Patients are rated on each of the 21 items on a scale of 0-6. Total scores are computed by adding up the scores of each individual item, with a total score ranging from 0-126. Higher scores reflect higher functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale | 71.8 (18.5) | 71.4 (15.6)

7. Secondary Outcome: Calgary Depression Scale for Schizophrenia (CDSS)
Description: Baseline scores on the Calgary Depression Scale for Schizophrenia (CDSS). Total CDSS scores range from 0-27. The assessment is comprised of 9 questions covering the topics of Depression, Hopelessness, Self Depreciation, Guilty Ideas of Reference, Pathological Guilt, Morning Depression, Early Wakening, Suicide, Observed Depression. Each item is scored on a scale from 0-3 (0 = absent, 1 = mild, 2 = moderate, 3 = severe). The total score is computed by adding up the individual scores of each item. The higher the score, the more prominent the symptoms of depression are for the participant.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale | 2.8 (3.1) | 3.4 (3.1)

8. Secondary Outcome: Clinical Global Impression (CGI)
Description: Considering you total clinical experience with this patient population, how mentally ill is the patient at this time?
  1=Normal, not at all, 2=Borderline mentally ill, 3=Mildy ill, 4=Moderately ill, 5=Markedly ill, 6=Severely ill, 7=Among the most extremely ill patients; a higher score indicates worse outcome
Time Frame: Weeks 0 and 8, and Month 6 after cognitive remediation completion
Population: 18 participants in each arm had baseline data available for analysis. At week 8, 17 participants in the D-cycloserine group and 15 in the placebo group had data available. At month 6, 6 participants in the D-cycloserine group and 4 in the placebo group had data available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
units on a scale
  Baseline | 3.78 (0.55) | 3.78 (0.73)
  Week 8: number analyzed (Participants) | 17 | 15
  Week 8 | 3.65 (0.61) | 3.73 (0.70)
  Month 6: number analyzed (Participants) | 6 | 4
  Month 6 | 4.00 (0.89) | 3.25 (0.50)

9. Secondary Outcome: Side Effects Checklist (SEC)
Description: Each side effect is entered as either yes or no for having had any severity of the side effect at each visit.
Time Frame: Weeks 0 - 8, and Month 6 after cognitive remediation completion
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | D-cycloserine | Placebo
Number analyzed (Participants) | 18 | 18
Participants
  Baseline : Bruising easily: Yes | 1 | 0
  Baseline : Bruising easily: No | 17 | 18
  Baseline : Rash: Yes | 0 | 3
  Baseline : Rash: No | 18 | 15
  Baseline : Urticaria (Hives, Itching): Yes | 1 | 4
  Baseline : Urticaria (Hives, Itching): No | 17 | 14
  Baseline : Blurred Vision: Yes | 0 | 2
  Baseline : Blurred Vision: No | 18 | 16
  Baseline : Sedation/Drowsiness: Yes | 4 | 7
  Baseline : Sedation/Drowsiness: No | 14 | 11
  Baseline : Restlessness: Yes | 6 | 6
  Baseline : Restlessness: No | 12 | 12
  Baseline : Insomnia: Yes | 3 | 6
  Baseline : Insomnia: No | 15 | 12
  Baseline : Malaise: Yes | 2 | 5
  Baseline : Malaise: No | 16 | 13
  Baseline : Stiffness: Yes | 5 | 5
  Baseline : Stiffness: No | 13 | 13
  Baseline : Tremor: Yes | 1 | 3
  Baseline : Tremor: No | 17 | 15
  Baseline : Dizziness: Yes | 3 | 2
  Baseline : Dizziness: No | 15 | 16
  Baseline : Headache: Yes | 2 | 4
  Baseline : Headache: No | 16 | 14
  Baseline : Fever: Yes | 0 | 0
  Baseline : Fever: No | 18 | 18
  Baseline : Sore Throat: Yes | 1 | 2
  Baseline : Sore Throat: No | 17 | 16
  Baseline : Dry Mouth: Yes | 5 | 9
  Baseline : Dry Mouth: No | 13 | 9
  Baseline : Hypersalivation: Yes | 1 | 1
  Baseline : Hypersalivation: No | 17 | 17
  Baseline : Enuresis: Yes | 0 | 2
  Baseline : Enuresis: No | 18 | 16
  Baseline : Constipation: Yes | 1 | 1
  Baseline : Constipation: No | 17 | 17
  Baseline : Diarrhea: Yes | 2 | 1
  Baseline : Diarrhea: No | 16 | 17
  Baseline : Anorexia: Yes | 0 | 4
  Baseline : Anorexia: No | 18 | 14
  Baseline : Nausea: Yes | 0 | 2
  Baseline : Nausea: No | 18 | 16
  Baseline : Vomiting: Yes | 0 | 2
  Baseline : Vomiting: No | 18 | 16
  Baseline : Menstrual Irregularities: Yes | 0 | 0
  Baseline : Menstrual Irregularities: No | 18 | 18
  Baseline : Breast Tenderness/Galactorrhea: Yes | 0 | 0
  Baseline : Breast Tenderness/Galactorrhea: No | 18 | 18
  Week 8 : Bruising easily: number analyzed (Participants) | 17 | 15
  Week 8 : Bruising easily: Yes | 0 | 0
  Week 8 : Bruising easily: No | 17 | 15
  Week 8 : Rash: number analyzed (Participants) | 17 | 15
  Week 8 : Rash: Yes | 2 | 1
  Week 8 : Rash: No | 15 | 14
  Week 8 : Urticaria (Hives, Itching): number analyzed (Participants) | 17 | 15
  Week 8 : Urticaria (Hives, Itching): Yes | 2 | 3
  Week 8 : Urticaria (Hives, Itching): No | 15 | 12
  Week 8 : Blurred Vision: number analyzed (Participants) | 17 | 15
  Week 8 : Blurred Vision: Yes | 1 | 1
  Week 8 : Blurred Vision: No | 16 | 14
  Week 8 : Sedation/Drowsiness: number analyzed (Participants) | 17 | 15
  Week 8 : Sedation/Drowsiness: Yes | 3 | 3
  Week 8 : Sedation/Drowsiness: No | 14 | 12
  Week 8 : Restlessness: number analyzed (Participants) | 17 | 15
  Week 8 : Restlessness: Yes | 2 | 6
  Week 8 : Restlessness: No | 15 | 9
  Week 8 : Insomnia: number analyzed (Participants) | 17 | 15
  Week 8 : Insomnia: Yes | 4 | 3
  Week 8 : Insomnia: No | 13 | 12
  Week 8 : Malaise: number analyzed (Participants) | 17 | 15
  Week 8 : Malaise: Yes | 3 | 1
  Week 8 : Malaise: No | 14 | 14
  Week 8 : Stiffness: number analyzed (Participants) | 17 | 15
  Week 8 : Stiffness: Yes | 1 | 3
  Week 8 : Stiffness: No | 16 | 12
  Week 8 : Tremor: number analyzed (Participants) | 17 | 15
  Week 8 : Tremor: Yes | 0 | 1
  Week 8 : Tremor: No | 17 | 14
  Week 8 : Dizziness: number analyzed (Participants) | 17 | 15
  Week 8 : Dizziness: Yes | 3 | 2
  Week 8 : Dizziness: No | 14 | 13
  Week 8 : Headache: number analyzed (Participants) | 17 | 15
  Week 8 : Headache: Yes | 0 | 2
  Week 8 : Headache: No | 17 | 13
  Week 8 : Fever: number analyzed (Participants) | 17 | 15
  Week 8 : Fever: Yes | 0 | 0
  Week 8 : Fever: No | 17 | 15
  Week 8 : Sore Throat: number analyzed (Participants) | 17 | 15
  Week 8 : Sore Throat: Yes | 0 | 2
  Week 8 : Sore Throat: No | 17 | 13
  Week 8 : Dry Mouth: number analyzed (Participants) | 17 | 15
  Week 8 : Dry Mouth: Yes | 3 | 5
  Week 8 : Dry Mouth: No | 14 | 10
  Week 8 : Hypersalivation: number analyzed (Participants) | 17 | 15
  Week 8 : Hypersalivation: Yes | 1 | 1
  Week 8 : Hypersalivation: No | 16 | 14
  Week 8 : Enuresis: number analyzed (Participants) | 17 | 15
  Week 8 : Enuresis: Yes | 0 | 1
  Week 8 : Enuresis: No | 17 | 14
  Week 8 : Constipation: number analyzed (Participants) | 17 | 15
  Week 8 : Constipation: Yes | 1 | 0
  Week 8 : Constipation: No | 16 | 15
  Week 8 : Diarrhea: number analyzed (Participants) | 17 | 15
  Week 8 : Diarrhea: Yes | 1 | 2
  Week 8 : Diarrhea: No | 16 | 13
  Week 8 : Anorexia: number analyzed (Participants) | 17 | 15
  Week 8 : Anorexia: Yes | 2 | 1
  Week 8 : Anorexia: No | 15 | 14
  Week 8 : Nausea: number analyzed (Participants) | 17 | 15
  Week 8 : Nausea: Yes | 0 | 1
  Week 8 : Nausea: No | 17 | 14
  Week 8 : Vomiting: number analyzed (Participants) | 17 | 15
  Week 8 : Vomiting: Yes | 0 | 0
  Week 8 : Vomiting: No | 17 | 15
  Week 8 : Menstrual Irregularities: number analyzed (Participants) | 17 | 15
  Week 8 : Menstrual Irregularities: Yes | 0 | 0
  Week 8 : Menstrual Irregularities: No | 17 | 15
  Week 8 : Breast Tenderness/Galactorrhea: number analyzed (Participants) | 17 | 15
  Week 8 : Breast Tenderness/Galactorrhea: Yes | 0 | 0
  Week 8 : Breast Tenderness/Galactorrhea: No | 17 | 15
  Month 6 : Bruising easily: number analyzed (Participants) | 6 | 4
  Month 6 : Bruising easily: Yes | 1 | 0
  Month 6 : Bruising easily: No | 5 | 4
  Month 6 : Rash: number analyzed (Participants) | 6 | 4
  Month 6 : Rash: Yes | 0 | 0
  Month 6 : Rash: No | 6 | 4
  Month 6 : Urticaria (Hives, Itching): number analyzed (Participants) | 6 | 4
  Month 6 : Urticaria (Hives, Itching): Yes | 0 | 1
  Month 6 : Urticaria (Hives, Itching): No | 6 | 3
  Month 6 : Blurred Vision: number analyzed (Participants) | 6 | 4
  Month 6 : Blurred Vision: Yes | 0 | 0
  Month 6 : Blurred Vision: No | 6 | 4
  Month 6 : Sedation/Drowsiness: number analyzed (Participants) | 6 | 4
  Month 6 : Sedation/Drowsiness: Yes | 1 | 2
  Month 6 : Sedation/Drowsiness: No | 5 | 2
  Month 6 : Restlessness: number analyzed (Participants) | 6 | 4
  Month 6 : Restlessness: Yes | 2 | 0
  Month 6 : Restlessness: No | 4 | 4
  Month 6 : Insomnia: number analyzed (Participants) | 6 | 4
  Month 6 : Insomnia: Yes | 1 | 0
  Month 6 : Insomnia: No | 5 | 4
  Month 6 : Malaise: number analyzed (Participants) | 6 | 4
  Month 6 : Malaise: Yes | 0 | 0
  Month 6 : Malaise: No | 6 | 4
  Month 6 : Stiffness: number analyzed (Participants) | 6 | 4
  Month 6 : Stiffness: Yes | 0 | 1
  Month 6 : Stiffness: No | 6 | 3
  Month 6 : Tremor: number analyzed (Participants) | 6 | 4
  Month 6 : Tremor: Yes | 0 | 1
  Month 6 : Tremor: No | 6 | 3
  Month 6 : Dizziness: number analyzed (Participants) | 6 | 4
  Month 6 : Dizziness: Yes | 1 | 1
  Month 6 : Dizziness: No | 5 | 3
  Month 6 : Headache: number analyzed (Participants) | 6 | 4
  Month 6 : Headache: Yes | 0 | 2
  Month 6 : Headache: No | 6 | 2
  Month 6 : Fever: number analyzed (Participants) | 6 | 4
  Month 6 : Fever: Yes | 0 | 0
  Month 6 : Fever: No | 6 | 4
  Month 6 : Sore Throat: number analyzed (Participants) | 6 | 4
  Month 6 : Sore Throat: Yes | 1 | 0
  Month 6 : Sore Throat: No | 5 | 4
  Month 6 : Dry Mouth: number analyzed (Participants) | 6 | 4
  Month 6 : Dry Mouth: Yes | 2 | 0
  Month 6 : Dry Mouth: No | 4 | 4
  Month 6 : Hypersalivation: number analyzed (Participants) | 6 | 4
  Month 6 : Hypersalivation: Yes | 2 | 0
  Month 6 : Hypersalivation: No | 4 | 4
  Month 6 : Enuresis: number analyzed (Participants) | 6 | 4
  Month 6 : Enuresis: Yes | 0 | 0
  Month 6 : Enuresis: No | 6 | 4
  Month 6 : Constipation: number analyzed (Participants) | 6 | 4
  Month 6 : Constipation: Yes | 0 | 1
  Month 6 : Constipation: No | 6 | 3
  Month 6 : Diarrhea: number analyzed (Participants) | 6 | 4
  Month 6 : Diarrhea: Yes | 2 | 1
  Month 6 : Diarrhea: No | 4 | 3
  Month 6 : Anorexia: number analyzed (Participants) | 6 | 4
  Month 6 : Anorexia: Yes | 1 | 0
  Month 6 : Anorexia: No | 5 | 4
  Month 6 : Nausea: number analyzed (Participants) | 6 | 4
  Month 6 : Nausea: Yes | 1 | 1
  Month 6 : Nausea: No | 5 | 3
  Month 6 : Vomiting: number analyzed (Participants) | 6 | 4
  Month 6 : Vomiting: Yes | 1 | 0
  Month 6 : Vomiting: No | 5 | 4
  Month 6 : Menstrual Irregularities: number analyzed (Participants) | 6 | 4
  Month 6 : Menstrual Irregularities: Yes | 0 | 0
  Month 6 : Menstrual Irregularities: No | 6 | 4
  Month 6 : Breast Tenderness/Galactorrhea: number analyzed (Participants) | 6 | 4
  Month 6 : Breast Tenderness/Galactorrhea: Yes | 0 | 0
  Month 6 : Breast Tenderness/Galactorrhea: No | 6 | 4

ADVERSE EVENTS:
Arm/Group | D-cycloserine | Placebo
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/18
Other Adverse Events (participants affected / at risk) | 17/18 | 13/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=18) | Placebo (N=18)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) — Patient was hospitalized due to worsening psychiatric symptoms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-cycloserine (N=18) | Placebo (N=18)
Bradycardia (Cardiac disorders) | 4 (8) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Drowsiness (General disorders) | 2 (2) | 0 (0)
Hypertension (Cardiac disorders) | 14 (32) | 13 (22)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 8 (15) | 6 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No